CLINICAL TRIAL: NCT03313804
Title: Priming Immunotherapy in Advanced Disease With Radiation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: John L. Villano, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, John L. Villano, MD, PhD, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17-MULTI-20-PMC
Record Dates: First submitted 2017-09-29; First posted 2017-10-18 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Non-small Cell Lung Cancer; Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck | interventions — Immune Checkpoint Inhibitors; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Immune Checkpoint Inhibitor + Radiation (Experimental): Immune checkpoint inhibitor (Nivolumab OR Pembrolizumab OR Atezolizumab) PLUS Radiation Therapy (Stereotactic Body Radiation Therapy OR fractionated radiation therapy)
  Interventions: Drug: Immune checkpoint inhibitor; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Immune checkpoint inhibitor — Standard of care immune checkpoint inhibitor
Radiation: Radiation Therapy — Stereotactic Body Radiation Therapy OR Fractionated radiation therapy

SUMMARY:
This study proposes to treat metastatic non-small cell lung cancer (NSCLC) and head/neck squamous cell cancer (HNSCC) patients who are already initiating an immune checkpoint inhibitor (such as Nivolumab, Atezolizumab or Pembrolizumab) for disease treatment as per FDA approved guidelines. In these patients we will deliver a short-course radiation to a single systemic (non-CNS) site within 14 days of receiving the first dose of immune checkpoint inhibitors. This sequence allows radiation to release tumor antigens from immune inaccessible areas such as necrotic tumor or low perfusion to provide a robust anti-tumor immune response with immune checkpoint inhibitors.

The primary objective is to assess six-month progression free survival (PFS) compared to historical control.

DETAILED DESCRIPTION:
Subjects with front-line or relapsed NSCLC or relapsed HNSCC who are intended to receive standard of care immune checkpoint inhibitors without a contraindication to Stereotactic Body Radiation Therapy (SBRT) to a single cancer deposit greater than 1 cm (metastasis or primary cancer) will be enrolled. Subjects will receive standard of care (SOC) immune checkpoint inhibitors and within 2 weeks of initiation, and will receive either:

* SBRT to target to achieve Biological Equivalent Dose (BED) > 100 Gy OR
* 30 Gy fractionated radiation therapy (RT) delivered as a 3 dimensional (3-D) dose.

The lesion choice will be made by the treating radiation oncologist and will be directed to a single malignant focus (non-CNS) that measures ≥ 1 cm. Essentially, the goals of both techniques are the same but SBRT is reserved for lesions that are readily encompassed by a single field with large RT fractions in which dose-limiting organs are within safe limits.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven advanced or metastatic non-small cell lung cancer or squamous cell carcinoma head and neck with tumor at least 1 cm in size.
2. Eligible for treatment with radiation therapy.
3. Prior treatment: chemotherapy or radiotherapy or surgery.

   1. Prior chemotherapy or radiation must have concluded ≥ 21 days prior to the start of study treatment.
   2. No limit is placed on prior systemic treatment, but subjects must be eligible for immune checkpoint inhibitors therapy, for an FDA approved indication.
   3. No major surgery within 14 days of start of study treatment.
4. No previous or concurrent malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease free for the past 3 years.
5. Age ≥ 18 years.
6. Life expectancy ≥ 3 months.
7. Required initial laboratory values:

   1. Absolute neutrophil count ≥ 1,000/mm3
   2. Platelets ≥ 100,000/mm3
   3. Total bilirubin ≤ 1.5 x ULN
   4. AST and ALT if no hepatic metastasis ≤ 2.5 times x ULN
   5. AST and ALT with hepatic metastasis ≤ 5 x ULN
   6. Creatinine ≤ 1.5 x ULN and Requires CrCl ≥ 60ml/min (per 24-hour urine collection or calculated according to the Cockcroft-Gault formula)
8. Non pregnant and non-nursing women. Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment. Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation. Subjects should use adequate birth control for at least 3 months after the last administration of immune checkpoint inhibitors.
9. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Active clinically serious infection > CTCAE Grade 2.
2. Serious non-healing wound, ulcer or bone fracture.
3. Prior treatment with immune checkpoint inhibitors.
4. Ineligible for immune checkpoint inhibitors based on package insert of the chosen immune checkpoint inhibitor (e.g., uncontrolled immunologic disorders, active hepatitis, active colitis, active pneumonitis, uncontrolled/active hormone gland problems - including thyroid, pituitary, adrenal glands and pancreas).
5. Major surgical procedure (including craniotomy and open brain biopsy) or significant traumatic injury within 14 days prior to registration or those patients who receive a non-CNS minor surgical procedures (e.g. core biopsy or fine needle aspiration) within 3 days prior to registration. There is no waiting period for central line placement. There is a 7-day window for recovery prior to registration for patients who underwent stereotactic biopsy of the brain.
6. Participants may not have uncontrolled inter-current illness. This includes, but is not limited to: ongoing or active infection; symptomatic congestive heart failure (NYHA class III or IV); unstable angina pectoris or new onset angina that began within the last 3 months; cardiac ventricular arrhythmias requiring anti-arrhythmic therapy; or thrombotic/embolic events such as cerebrovascular accident, including transient ischemic attacks within the past 6 months. Uncontrolled hypertension defined as systolic blood pressure >150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management. Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C. Known Grade 3 or 4 neurotoxicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2026-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John Villano, MD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 76 participants were enrolled but 1 participant never received treatment and therefore was not counted in the on treatment (started) number.
Period: Treatment
Arm/Group | Immune Checkpoint Inhibitor + Radiation
Started | 75
Completed | 68
Not Completed | 7
Not completed — Death | 5
Not completed — still on treatment | 2
Period: Follow Up
Arm/Group | Immune Checkpoint Inhibitor + Radiation
Started | 68
Completed | 65
Not Completed | 3
Not completed — still on follow up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Immune Checkpoint Inhibitor + Radiation
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.51 (8.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 73
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 64
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 75

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Alive and Without Progression
Description: Progression-free survival will be calculated as a rate, time from enrollment in the study to progression at 6-months post enrollment.
Time Frame: 6-months post enrollment
Measure: Number; unit: proportion of participants
Arm/Group | Immune Checkpoint Inhibitor + Radiation
Number analyzed (Participants) | 67
proportion of participants | .66

2. Secondary Outcome: Percentage of (Programmed Death) PD-1+ CD4+ T (Helper) Cells and PD-1+ CD8+ T (Cytotoxic) Cells Prior to Treatment Versus With Concurrent Treatment.
Time Frame: Assessed at specified points--1) prior to each cycle of therapy for 4 cycles (one cycle equals 6 weeks) 2) at disease progression (date first progression post-randomization, assessed up to 3 years) 3) when participant is off-study, assessed up to 3 years
Reporting Status: Not Posted

3. Secondary Outcome: Percentage of CD8+ T-cells That Are Gamma-interferon Positive During Treatment.
Time Frame: as for outcome 2
Reporting Status: Not Posted

4. Secondary Outcome: Percentage PD-L1+ CD4+ and PD-L1+ CD8+ T-cell Expression Differences During Treatment
Time Frame: as for outcome 2
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 years
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for AE reporting
Arm/Group | Immune Checkpoint Inhibitor + Radiation
All-Cause Mortality (participants affected / at risk) | 30/75
Serious Adverse Events (participants affected / at risk) | 45/75
Other Adverse Events (participants affected / at risk) | 72/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Immune Checkpoint Inhibitor + Radiation (N=75)
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Lymphocyte count decreased (Investigations) | 17
Alkaline phosphatase increased (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Creatinine increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Fatigue (General disorders) | 1
Edema limbs (General disorders) | 1
Edema face (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Disease progression (General disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Oral hemorrhage (Gastrointestinal disorders) | 2
Anal hemorrhage (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Anemia (Blood and lymphatic system disorders) | 3
Leukocytosis (Blood and lymphatic system disorders) | 1
Other (Blood and lymphatic system disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Other (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Headache (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Muscle weakness right-sided (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Other (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Joint infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Confusion (Psychiatric disorders) | 2
Delirium (Psychiatric disorders) | 1
Hypotension (Vascular disorders) | 3
Hypertension (Vascular disorders) | 1
Superior vena cava syndrome (Vascular disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Other (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Immune Checkpoint Inhibitor + Radiation (N=75)
Hyponatremia (Metabolism and nutrition disorders) | 28
Hypoalbuminemia (Metabolism and nutrition disorders) | 24
Hypokalemia (Metabolism and nutrition disorders) | 14
Hyperglycemia (Metabolism and nutrition disorders) | 16
Hyperkalemia (Metabolism and nutrition disorders) | 13
Hypocalcemia (Metabolism and nutrition disorders) | 13
Hypomagnesemia (Metabolism and nutrition disorders) | 8
Hypercalcemia (Metabolism and nutrition disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 5
Hypoglycemia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Other (Metabolism and nutrition disorders) | 1
Lymphocyte count decreased (Investigations) | 26
Alkaline phosphatase increased (Investigations) | 19
Alanine aminotransferase increased (Investigations) | 11
Aspartate aminotransferase increased (Investigations) | 10
Thyroid stimulating hormone increased (Investigations) | 8
Creatinine increased (Investigations) | 6
Platelet count decreased (Investigations) | 6
White blood cell decreased (Investigations) | 5
Neutrophil count decreased (Investigations) | 1
Hemoglobin increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Cardiac troponin T increased (Investigations) | 1
CPK increased (Investigations) | 1
Other (Investigations) | 1
Lymphocyte count increased (Investigations) | 1
Weight gain (Investigations) | 1
Weight loss (Investigations) | 1
Urine output decreased (Investigations) | 1
Fatigue (General disorders) | 27
Edema limbs (General disorders) | 8
Edema face (General disorders) | 5
Pain (General disorders) | 5
Fever (General disorders) | 3
Gait disturbance (General disorders) | 3
Neck edema (General disorders) | 3
Non-cardiac chest pain (General disorders) | 2
Chills (General disorders) | 2
Other (General disorders) | 1
Facial pain (General disorders) | 1
Localized edema (General disorders) | 1
Nausea (Gastrointestinal disorders) | 13
Diarrhea (Gastrointestinal disorders) | 10
Dysphagia (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 5
Dry mouth (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Oral hemorrhage (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 3
Mucositis oral (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Other (Gastrointestinal disorders) | 1
Oral dysesthesia (Gastrointestinal disorders) | 1
Small intestinal mucositis (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 3
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1
Other (Musculoskeletal and connective tissue disorders) | 1
Head soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 18
Eosinophilia (Blood and lymphatic system disorders) | 6
Leukocytosis (Blood and lymphatic system disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13
Other (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 1
Headache (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 2
Peripheral motor neuropathy (Nervous system disorders) | 2
Muscle weakness right-sided (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Sinusitis (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 3
Eye infection (Infections and infestations) | 2
Other (Infections and infestations) | 1
Skin infection (Infections and infestations) | 2
Lung infection (Infections and infestations) | 1
Papulopustular rash (Infections and infestations) | 2
Hepatitis viral (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Thrush (Infections and infestations) | 1
Confusion (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 5
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Hallucinations (Psychiatric disorders) | 1
Hypotension (Vascular disorders) | 3
Hypertension (Vascular disorders) | 3
Hot flashes (Vascular disorders) | 1
Hypothyroidism (Endocrine disorders) | 6
Hyperthyroidism (Endocrine disorders) | 2
Other (Endocrine disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 2
Other (Ear and labyrinth disorders) | 2
Bruising (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 2
Other (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Wound complication (Injury, poisoning and procedural complications) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 1
Dysuria (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 1
Dry eye (Eye disorders) | 2
Other (Eye disorders) | 1
Genital edema (Reproductive system and breast disorders) | 2
Pelvic pain (Reproductive system and breast disorders) | 2
Other (Immune system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-06): https://cdn.clinicaltrials.gov/large-docs/04/NCT03313804/Prot_SAP_000.pdf